CLINICAL TRIAL: NCT03296033
Title: Evaluation of Residual Anti-Xa Activity As A Function Of Time Following The Last Treatment Dose of Enoxaparin In Patients Presenting For Elective Surgery
Brief Title: Residual Anti-Xa Activity After Last Treatment Dose of Enoxaparin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: enrollment proved to be a challenge due to the changing of the guidelines for bridging off the new anticoagulants that are being prescribed
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00044503
Record Dates: First submitted 2017-07-06; First posted 2017-09-28 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Anticoagulants and Bleeding Disorders; Surgery; Regional Anesthesia Morbidity
Keywords: enoxaparin; thromboembolism; coagulation; factor Xa
MeSH Terms: conditions — Hemostatic Disorders; Thromboembolism; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: After consenting to the study, patients will be randomized to one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24 Hours group (Active Comparator): Group one will be instructed to administer their last dose of enoxaparin at 07:00 in the morning on the day prior to their scheduled surgery date. This will mean that patients who have their surgery scheduled for 07:00 the following day will be 24-hours removed from their last dose. Patients presenting for surgery later in the day would be slightly farther removed from their last dose, however this is currently considered normal clinical practice.
  Interventions: Drug: Enoxaparin
- 36 Hours Group (Experimental): Group 2 will be instructed to administer their last dose of enoxaparin at 19:00 in the evening two days prior to their scheduled surgery date. Patients presenting for surgery at 07:00 two days later will be 36-hours removed from their last dose. Patients presenting for surgery later in the day would be slightly farther removed from their last dose, but again this mimics normal clinical practice in which the timing of the last dose of self-administered enoxaparin is not routinely adjusted based on the scheduled surgical start time.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — The intervention is the implementation of a 36-hour time period from the last dose of treatment dose Enoxaparin to the blood sampling for anti-Xa testing.
  Other Names: Lovenox
  Arms: 36 Hours Group
Drug: Enoxaparin — This is the historical control arm. 24 hours removed from their last dose (time period from the last dose of treatment dose Enoxaparin to the blood sampling for anti-Xa testing)
  Other Names: Lovenox
  Arms: 24 Hours group

SUMMARY:
The main objective of this study is to determine the time interval following the last treatment dose of enoxaparin at which the amount of anti-Xa level activity is reliably less than 0.2 international unit per milliliter (IU/mL) in patients presenting for elective surgery.

DETAILED DESCRIPTION:
Enoxaparin is a factor Xa inhibitor commonly used for both prophylaxis against and treatment of thromboembolism. It is also frequently used off-label as a perioperative bridge for patients that are chronically anticoagulated prior to surgery, such as those taking Warfarin. It is an attractive option for perioperative use secondary to its predictable pharmacologic profile and the lack of recommended routine blood monitoring. Therefore, it is common to encounter a patient who has recently received a treatment dose of Enoxaparin prior to presenting for surgery. For these patients, and those on other anticoagulant medications, published guidelines have been developed to help guide clinical decision-making when the anesthetic/analgesic plan includes regional anesthesia.1 Currently, these guidelines recommend that a minimum of 24-hours should elapse following the last treatment dose of Enoxaparin before a neuraxial procedure is performed. However, a recently completed quality improvement project conducted at Wake Forest Baptist Medical Center found that almost 60% of patients presenting for surgery while on treatment dose enoxaparin still had significant anticoagulant activity 24-hours following their last dose, as demonstrated by anti-Xa level assay testing. Given that the risk of epidural hematoma formation is increased in the setting of abnormal coagulation parameters, the significance of this finding is that the risk of bleeding complications following a neuraxial procedure may still be increased 24-hours after the last treatment dose of enoxaparin.

While the routine use of anti-Xa level testing may be a viable option to determine when residual enoxaparin activity is present before proceeding with a neuraxial procedure on a patient-by-patient basis, it is not universally available at all hospitals. Therefore, it is important to determine the time interval following the last enoxaparin dose at which the likelihood that a clinically relevant amount of residual anti-Xa level activity no longer persists, so that providers can confidently proceed with a neuraxial procedure when anti-Xa level testing is not available.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients need:

* to be on treatment dose (1mg/kg twice daily or 1.5mg/kg daily) enoxaparin at the time of presentation for elective surgery
* and must be able to accurately report the timing of their last dose and the administered dosage.
* Patients must also be between the ages of 18-100 years of age
* and must be able to give written consent to participate.

Exclusion Criteria:

* Patients with severe renal insufficiency (creatinine clearance <30ml/min) will be excluded from the study, as the elimination of enoxaparin is known to be affected in this patient population.
* Pregnant patients will also be excluded, as the elimination and metabolism of enoxaparin is known to be altered in this patient population, and dose adjustments are recommended if treatment dose enoxaparin is used during pregnancy.
* Patients who are receiving enoxaparin as a bridge from another anti-Xa inhibiting medication will be excluded as this could unpredictably affect the results of anti-Xa testing. These medications include: Apixaban, Edoxaban, Fondaparinux, and Xarelto.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Henshaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horlocker TT, Wedel DJ, Rowlingson JC, Enneking FK, Kopp SL, Benzon HT, Brown DL, Heit JA, Mulroy MF, Rosenquist RW, Tryba M, Yuan CS. Regional anesthesia in the patient receiving antithrombotic or thrombolytic therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Third Edition). Reg Anesth Pain Med. 2010 Jan-Feb;35(1):64-101. doi: 10.1097/aap.0b013e3181c15c70. PMID 20052816
- [Result] Henshaw DS, Turner JD, Forest DJ, Thompson GR, Weller RS. Residual Enoxaparin Activity, Anti-Xa Levels, and Concerns About the American Society of Regional Anesthesia and Pain Medicine Anticoagulation Guidelines. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):432-436. doi: 10.1097/AAP.0000000000000617. PMID 28492441
- [Derived] Henshaw DS, Edwards CJ, Dobson SW, Jaffe D, Turner JD, Reynolds JW, Thompson GR, Russell G, Weller R. Evaluating residual anti-Xa levels following discontinuation of treatment-dose enoxaparin in patients presenting for elective surgery: a prospective observational trial. Reg Anesth Pain Med. 2024 Feb 5;49(2):94-101. doi: 10.1136/rapm-2023-104571. PMID 37280083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 24 Hours Group | 36 Hours Group
Started | 60 | 62
Completed | 51 | 52
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Population: Baseline characteristics only collected for subjects who completed
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 Hours Group | 36 Hours Group | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (12.1) | 65.5 (13.5) | 64.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 30 | 29 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Residual Anti-Xa Activity Levels Following Last Treatment Dose of Enoxaparin
Description: Anti-Xa level activity will be measured in both groups using a chromogenic assay and a hybrid curve calibrated to both heparin and enoxaparin.
Time Frame: Time Frame: 24 hours or 36 hours (based on randomization) after the last treatment dose of enoxaparin. Actual lab draw will vary, as planned, given surgical arrival time.
Population: The two groups/arms were compared here as this outcome was considered part of the demographic group comparison, much like age or sex.
Measure: Mean (Standard Deviation); unit: international units per mililiter IU/ mL
Arm/Group | 24 Hours Group | 36 Hours Group
Number analyzed (Participants) | 51 | 52
international units per mililiter IU/ mL | .23 (.17) | .11 (.06)

2. Primary Outcome: Time Point at Which Anti-Xa Activity is Lower Than 0.2 International Unit Per Milliliter (IU/mL) Using Modeling
Description: The randomization of patients to either the 24-hour group or the 36-hour group will allow for modeling, which will generate a prediction of the time point at which the level of anti-Xa activity can reliably be assumed to be lower than 0.2 IU/mL.
Time Frame: as for outcome 1
Population: On note: Arms/Groups were combined together for analysis purposes and results are reported in this same fashion. The approach was planned apriori. A comparison between the two groups in regard to this primary outcome was neither planned nor performed. Including both arms/groups in a single data set allowed for logistical regression, which was utilized to determine the overall estimate of time until residual anti-Xa level activity reliably fell below 0.2IU/mL).
Measure: Mean (95% Confidence Interval); unit: time in hours
Groups:
- Both Together: Both 24hr and 36hr arms analyzed together
Arm/Group | Both Together
Number analyzed (Participants) | 103
time in hours | 31.4 [25.0 to 31.5]

3. Secondary Outcome: Relationship Between Anti-Xa Levels and Patient Age
Description: Analyze and determine the best-fit function (beta and standard error) for anti-Xa activity level activity (IU/mL) to determine if there is a significant association between anti-Xa activity at the time of presentation and patient age (years).
  Individual patient characteristics were assessed to determine their impact on the odds of success, defined as an anti-Xa level of <0.2IU/mL. Patient characteristics assessed included age, sex, renal function (calculated by Cockcroft-Gault and modified Cockcroft-Gault formulae), and body mass index (BMI), the latter of which was assessed post-hoc.
  Odds ratios were calculated with both groups combined, as time from last dose varied and even overlapped between groups, which was expected/anticipated as part of the study design. All patient characteristics were analyzed using three separate time intervals from last dose (<24-hours, 24-hours through 35.9-hours, and >36-hours).
Time Frame: Anti-Xa levels were measured at the time of presentation for surgery. Age was collected at the time of enrollment.
Population: All patients were included in a single analysis (planned priori) to assess the association between age and residual anti-Xa level activity at the time of presentation, which reflects time from last dose. Data for the association between anti-Xa level activity and age is shown below. Note "number" represents Odds Ratio (OR) with corresponding 95% CI. This outcome was planned to be analyzed as one arm per protocol.
Measure: Number (95% Confidence Interval); unit: Odds Ratio (Per 5-year change)
Arm/Group | Both Together
Number analyzed (Participants) | 103
Odds Ratio (Per 5-year change) | 0.99 [0.83 to 1.18]

4. Secondary Outcome: Relationship Between Anti-Xa Levels and Patients Gender (Sex)
Description: Analyze and determine the best-fit function (beta and standard error) for anti-Xa activity level activity (IU/mL) to determine if there is a significant association between anti-Xa activity at the time of presentation and (gender= male or female).
  Individual patient characteristics were assessed to determine their impact on the odds of success, defined as an anti-Xa level of <0.2IU/mL. Patient characteristics assessed included age, sex, renal function (calculated by Cockcroft-Gault and modified Cockcroft-Gault formulae), and body mass index (BMI), the latter of which was assessed post-hoc.
  Odds ratios were calculated with both groups combined, as time from last dose varied and even overlapped between groups, which was expected/anticipated as part of the study design. All patient characteristics were analyzed using three separate time intervals from last dose (<24-hours, 24-hours through 35.9-hours, and >36-hours).
Time Frame: Anti-Xa levels were measured at the time of presentation for surgery. Gender was collected at the time of enrollment.
Population: All patients were included in a single analysis (planned priori) to assess the association between gender (sex) and residual anti-Xa level activity at the time of presentation, which reflects time from last dose. Data for the association between anti-Xa level activity and gender (sex) is shown below. Note "number" represents Odds Ratio (OR) with corresponding 95% CI. This outcome was planned to be analyzed as one arm per protocol.
Measure: Number (95% Confidence Interval); unit: Odds Ratio (OR) female vs male
Arm/Group | Both Together
Number analyzed (Participants) | 103
Odds Ratio (OR) female vs male | 0.91 [0.38 to 2.20]

5. Other Pre Specified Outcome: Relationship Between Anti-Xa Levels and Patient Renal Function
Description: Analyze and determine the best-fit function (beta and standard error) for anti-Xa activity level activity (IU/mL) to determine if there is a significant association between anti-Xa activity at the time of presentation and renal function.
  Individual patient characteristics were assessed to determine their impact on the odds of success, defined as an anti-Xa level of <0.2IU/mL. Patient characteristics assessed included age, sex, renal function (calculated by Cockcroft-Gault and modified Cockcroft-Gault formulae), and body mass index (BMI), the latter of which was assessed post-hoc.
  Odds ratios were calculated with both groups combined, as time from last dose varied and even overlapped between groups, which was expected/anticipated as part of the study design. All patient characteristics were analyzed using three separate time intervals from last dose (<24-hours, 24-hours through 35.9-hours, and >36-hours).
Time Frame: Anti-Xa levels were measured at the time of presentation for surgery as was glomerular filtration rates, which were used to calculate creatinine clearance.
Population: All patients were included in a single analysis (planned priori) to assess the association between renal function and residual anti-Xa level activity at the time of presentation, which reflects time from last dose. Data for the association between anti-Xa level activity and renal function are shown below. Note "number" represents Odds Ratio (OR) with corresponding 95% CI. This outcome was planned to be analyzed as one arm per protocol.
Measure: Number (95% Confidence Interval); unit: Odds Ratio Modified Cockcroft-Gault
Groups:
- All Together: Both 24hr and 36hr arms analyzed together
Arm/Group | All Together
Number analyzed (Participants) | 103
Odds Ratio Modified Cockcroft-Gault
  Using Cockcroft-Gault Forumula to estimate renal function | 0.97 [0.89 to 1.06]
  Using modified Cockcroft-Gault formula to estimate renal function | 0.98 [0.86 to 1.11]

ADVERSE EVENTS:
Time Frame: From baseline through 36 hours
Arm/Group | 24 Hours Group | 36 Hours Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03296033/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03296033/ICF_000.pdf